CLINICAL TRIAL: NCT06382441
Title: A Pilot Study of "a Home-based and Group-based Tele-exercise Program for Breast Cancer Survivors: a Randomized Controlled Trial"
Brief Title: A Tele-exercise Program for Breast Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Principal Investigator, Gao Yang, Associate Professor, Hong Kong Baptist University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KC/KE-23-0122/ER-4
Record Dates: First submitted 2024-03-05; First posted 2024-04-24 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Behavior, Health
Keywords: tele-exercise; breast cancer survivors; randomized controlled trial
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tele-excercise (Experimental): In Group A (intervention), the 12 participants will form 2 groups (6 participants per group) according to their individual exercise intensity levels determined prior to the intervention for each participant. Each group will receive online coach-supervised training sessions 3 times per week for 4 weeks (a total of 12 sessions), which will be delivered by a certified coach and an assistant (a student helper, major in sports and health). Each session will consist of warm-up, aerobic exercise, resistance exercise, stretching and cool-down, with exercise period progressively increasing from 30 minutes to 50 minutes and exercise intensity progressively increasing from low to moderate levels (Table 1). Lighter intensity may be adopted when there is a need (e.g., for those with severe conditions). Target heart rate during exercise will be monitored by a pulse oximeter. Cameras will be requested to be turned on all the time.
  Interventions: Behavioral: tele-exercise
- Control (No Intervention): Participants in Group B (active control) will receive an essay on exercise and health every week for four weeks (a total of 4 essays). Proposed topics include: 1) beneficial effects of exercise and recommended exercise for breast cancer survivors; 2) WHO's recommendations for physical activity; 3) exercise intensity; 4) principles of exercise.

INTERVENTIONS:
Behavioral: tele-exercise — It is a prospective and pilot study of RCT. It will be a pilot to test acceptability and feasibility of a two-armed tele-exercise RCT to mitigate symptoms and improve health for breast cancer survivors. In this study, outcome assessors and data analysts will be masked from the allocation results. The pilot will recruit 24 patients and randomly assign them to an intervention group (Group A) and an active control group (Group B). All participants in both groups will continue receiving usual care from the study hospital during the study period. Additionally, those in Group A (intervention) will receive the tele-exercise (12 home-based online training sessions + 4 psychological counselling sessions), while those in Group B (active control) will receive 4 essays on exercise and health. Outcome measurements will be repeatedly performed before and after the intervention.
  Arms: Tele-excercise

SUMMARY:
The research protocol outlines a pilot study for a home-based and group-based tele-exercise program designed for breast cancer survivors. The study is a randomized controlled trial (RCT) led by Dr. Yang Gao from Hong Kong Baptist University, with multiple other investigators from Kwong Wah Hospital and the university itself.

Breast cancer is identified as the most prevalent cancer among women globally and in Hong Kong. The document states that adjuvant therapies post-surgery, such as radiation and chemotherapy, can have both short-term and long-term side effects, which may affect the survivors' physical and mental health.

The study is based on evidence that physical activity levels often decrease after a breast cancer diagnosis and that exercise can mitigate the side effects of treatment, improving health and quality of life. The pilot aims to test the acceptability and feasibility of a 12-week tele-exercise program that combines psychological theories and behaviour change techniques, transitioning from supervised to unsupervised exercise to build sustainable exercise habits.

The study will enrol 24 patients, randomly assigning them to an intervention group or an active control group. The intervention group will receive 12 online training sessions plus 4 psychological counselling sessions, whereas the control group will receive educational essays on exercise and health.

The training sessions for the intervention group will include various exercises with increasing intensity and duration over the 4 weeks, monitored by a pulse oximeter to ensure exercises are done at the appropriate heart rate. The sessions will be led by qualified coaches, with Dr. Gao overseeing quality control.

DETAILED DESCRIPTION:
It is a prospective and pilot study of RCT. It will be a pilot to test the acceptability and feasibility of a two-armed tele-exercise RCT to mitigate symptoms and improve health for breast cancer survivors. In this study, outcome assessors and data analysts will be masked from the allocation results. The pilot will recruit 24 patients and randomly assign them to an intervention group (Group A) and an active control group (Group B). All participants in both groups will continue receiving usual care from the study hospital during the study period. Additionally, those in Group A (intervention) will receive the tele-exercise (12 home-based online training sessions + 4 psychological counselling sessions), while those in Group B (active control) will receive 4 essays on exercise and health. Outcome measurements will be repeatedly performed before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 40-64 years old;
* Within 6 weeks after completion of chemotherapy;
* Without severe anemia;
* Without cancer metastasis;
* Able to read and communicate in Cantonese or Mandarin;
* Smartphone users.

Exclusion Criteria:

* With any medical, physical and psychological conditions that may limit participation (e.g., uncontrolled severe cardiovascular disease, schizophrenia, severe neurological dysfunction, etc.).

Ages: 40 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Acceptability (quantitative) | baseline, 13 weeks
  Participants rated intervention regarding the aspects of satisfaction, enjoyment, perceptions of safety, difficulty, tolerability of treatment, adverse events using a 5-Liker questionnaire, mean score was used to assess, and higher score indicates greater acceptability.
Acceptability (qualitative) | baseline, 13 weeks
  Participants rated intervention regarding the aspects of satisfaction, enjoyment, perceptions of safety, difficulty, tolerability of treatment, adverse events by interviews.
Recruitment rate | baseline, 13 weeks
  The proportion of eligible participants who are enrolled at baseline of the study.
Retention rate | baseline, 13 weeks
  The proportion of enrolled participants who are present throughout the full length of the treatment.
Attendance rate | baseline, 13 weeks
  The proportion of total sessions offered to participants to the actual number of sessions participants attended.
Compliance rate | baseline, 13 weeks
  Participants' level of adherence to the content, frequency, duration, and coverage of the treatment as delivered by the research team. Assessed by percentage of participants who complied with intervention procedures.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | baseline, 13 weeks
  estimated by the 6-minute walk test, primary outcome of the main study
muscle strength | baseline, 13 weeks
  upper extremity muscle strength by the hand grip test and lower extremity muscle strength by the timed stand test
balance | baseline, 13 weeks
  Assessed using the Single Leg Stance Test. It is used to assess static postural and balance control and widely used in clinical settings to monitor neurological and musculoskeletal conditions.
% body fat | baseline, 13 weeks
  A Body Composition Analyzer (InBody 270)
skeletal muscle mass | baseline, 13 weeks
  A Body Composition Analyzer (InBody 270)
height | baseline, 13 weeks
  Measured using a portable stadiometer
Shoulder joint range of motion (ROM) of affected side | baseline, 13 weeks
  An arm goniometer will be used to measure shoulder joint ROM in forward flexion, internal rotation, external rotation, and abduction, following the Struyf and Meeus' recommendations to conduct the goniometric shoulder joint ROM measurements
Limb circumference and lymphedema | baseline, 13 weeks
  Arm circumference will be measured with a non-stretch tape at styloid and every 10 cm intervals from the ulnar styloid up to 40 cm distally 19. D Lymphedema will be defined as a more than 2 cm between-arm difference in arm circumference at any measurement point.
Health-related quality of life | baseline, 13 weeks
  Functional Assessment of Cancer Therapy - Breast (FACT-B) will be used. The total score of FACT-B ranged from 0 t o148. The higher the score, the better the quality of life.
Physical activity level (min/week) | baseline, 13 weeks
  International physical activity questionnaire (short version) was used to calculate physical activity level (min/week), higher scores mean a greater physical acitivity level.

CONTACTS AND LOCATIONS:
Overall Officials: Oi Kwan CHUN, Study Director — Dept of Surgery, KWH; Wai Wun Sara FUNG, Study Director — Dept of Surgery, KWH
Locations (2):
- Hong Kong (2):
  - Xiong Zhennan, Kowloon Tong, Kowloon
  - Yan SUN, Kowloon Tong, Kowloon

IPD SHARING:
Plan to Share IPD: No